CLINICAL TRIAL: NCT04091165
Title: Mobile APP Utilization for Enhanced Post-Operative Nutritional Recovery
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-19978
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: GI Cancer; Nutritional Deficiency
Keywords: food diary; malnutrition
MeSH Terms: conditions — Gastrointestinal Neoplasms; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Participants will be identified for inclusion by leaders of the GI Clinic after GI surgery has been scheduled. Upon consenting, participants will be instructed how to download and use the mobile phone application "My Plate Calorie Counter".
  Interventions: Other: My Plate Calorie Tracker

INTERVENTIONS:
Other: My Plate Calorie Tracker — My Plate Calorie Tracker is a user-friendly weight management, calorie record application, available for smart phone devices. Users have the option to input items manually (i.e., calories, carbohydrates, fats, and proteins), select from a list of popular food items, or scan barcodes on the food packaging. In addition to food entries, users can also enter daily water intake and physical activities. Once an account is created, data entered into the mobile application can be sync'd to the "My Plate Calorie Tracker" website.
  Other Names: mobile application

SUMMARY:
This study is to assess the usability and acceptability of a digital food consumption diary as part of the perioperative management of gastrointestinal oncology patients and to evaluate the impact of a digital food diary on adherence to dietician-recommended plan and on quality recovery, using a commercially available smart phone application.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastrointestinal (GI) cancers confirmed by tissue diagnosis and/or clinical presentation as judged by the treating physician
* Candidate for curative-intent surgery
* Participants will be eligible for participation regardless of degree of malnutrition (as determined at pre-operative dietary consultation)
* Own a smartphone with iOS or Android operating systems with WiFi or 3G/4G connection
* Willingness to download the Livestrong.com MyPlate Calorie Tracker onto a personal smart phone with assumption and responsibility for individual data usage, and creation of login for website data extraction
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Sufficient English language proficiency to execute study tasks

Exclusion Criteria:

* Participants with tube feeds and/or need for parenteral/enteral nutrition
* Participants not willing to download or utilize the commercially available weight monitoring application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery in the Moffitt GI Clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Usability of Smart Phone Application | Up to 3 months
  Usability of smart phone application will be captured by (1) number of days that entries have been made by the study participants and recorded as a percentage of the total number of days after discharge from the hospital (obtained from mobile application (2) number of meals recorded in the application per day (obtained from mobile application) and (3) Exit Questionnaire (6 questions of 12). The Exit Questionnaire includes a mixture of 5-point Likert-scale, yes or no, and open-ended items to assess usability. Questions on the 5 point scale use 1 as an indication of difficulty in using application and 5 would be ease of use.
Acceptability of Smart Phone Application | Up to 3 months
  Patient's acceptability of the mobile application to assist with postoperative nutrition goals will be captured by the Exit Questionnaire (6 questions of 12). The Exit Questionnaire includes a mixture of 5-point Likert-scale, yes or no, and open-ended items to assess acceptability. Questions on the 5 point scale use 1 as an indication of acceptability issues of the application and 5 would be acceptability.

SECONDARY OUTCOMES:
Adherence to Recommended Nutritional Plan | Up to 3 months
  Adherence to the participant's recommended nutritional plan will be calculated by participant's energy (caloric) intake over time, as recorded in the digital food diary, and compared to estimates of the optimum energy needs established by the dietician. Adherence will be reported as a percentage of estimated energy requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Hodul, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer & Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Allenson K, Turner K, Gonzalez BD, Gurd E, Zhu S, Misner N, Chin A, Adams M, Cooper L, Nguyen D, Naffouje S, Castillo DL, Kocab M, James B, Denbo J, Pimiento JM, Malafa M, Powers BD, Fleming JB, Anaya DA, Hodul PJ. Pilot trial of remote monitoring to prevent malnutrition after hepatopancreatobiliary surgery. BMC Nutr. 2021 Dec 9;7(1):82. doi: 10.1186/s40795-021-00487-3. PMID 34886909

DOCUMENTS (1):
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04091165/ICF_000.pdf